CLINICAL TRIAL: NCT07323043
Title: The Affiliated Lianyungang Hospital of Xuzhou Medical University
Brief Title: Comparison of Cough Response Between Tegilidine and Sufentanil as Pre-induction Agents in General Anesthesia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First People's Hospital of Lianyungang (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KY-20250815003-01
Record Dates: First submitted 2025-11-23; First posted 2026-01-07 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: General Anesthetic Drug Adverse Reaction
MeSH Terms: interventions — Sufentanil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tegilidine group (Experimental): Administer 20-50ug/kg of Tegilidine before induction of general anesthesia, and record the patient's coughing episodes 2 minutes after administration. Then proceed with anesthesia induction.
  Interventions: Drug: Tegilidine
- Sufentanil group (Active Comparator): Administer sufentanil 0.4 µg/kg before the induction of general anesthesia, and record the patient's coughing episodes 2 minutes after administration. Then proceed with anesthesia induction.
  Interventions: Drug: Sufentanil

INTERVENTIONS:
Drug: Tegilidine — Inject Tegilidine in the induction of general anesthesia
  Arms: Tegilidine group
Drug: Sufentanil — Inject Sufentanil in the induction of general anesthesia
  Arms: Sufentanil group

SUMMARY:
In patients undergoing general anesthesia with planned tracheal intubation , a prospective, randomized, controlled, double-blind study was conducted to record the occurrence of cough 2 minutes after injection of Sufentanil or tegilidine. The cough was graded based on the frequency and duration: Grade I, no cough; Grade II, a single mild cough; Grade III, multiple coughs with duration <1 second; Grade IV, continuous coughing with a duration >15 seconds.

DETAILED DESCRIPTION:
Using a computer-generated randomized number table, patients were divided into two groups: the experimental group receiving Tiliglitidine (T group) at 20-50ug/kg, and the control group receiving Sufentanil (S group) at 0.4 μg/kg. After patients arrived in the operating room, routine monitoring including non-invasive blood pressure, electrocardiogram, and oxygen saturation was performed, and intravenous access was established. Patients were oxygenated and given the study drug before anesthesia induction. No other drugs were administered to the patients before giving the study drug. During anesthesia induction, patients received intravenous injection of Tiliglitide or Sufentanil according to their group. The severity of coughing was graded based on the number of coughing episodes: graded by the number and duration of coughs: Grade I, no cough, breathing regular; Grade II, a single mild cough; Grade III, multiple coughs, lasting less than 15 seconds; Grade IV, continuous coughs, lasting more than 15 seconds.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 65 years, 18 ≤ BMI (kg/m²) ≤ 30;
2. ASA grade I ~ III;
3. Scheduled elective surgery under general anesthesia with tracheal intubation.

Exclusion Criteria:

1. Patients with chronic cough (cough lasting >8 weeks) or asthma;
2. Patients with a history of allergy to the drugs used during the study;
3. Patients with severe cardiovascular disease, intracranial lesions, eye lesions, or lung lesions.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2026-01-15 (Actual); Primary Completion 2026-05-16 (Estimated); Study Completion 2026-06-16 (Estimated)

PRIMARY OUTCOMES:
Incidence of choking cough response | 2 minutes after administration
  Two minutes after administration of the study drugs (Tegilidine/Sufentanil), any clear coughing action is considered an 'occurrence'.

SECONDARY OUTCOMES:
Grading of choking and coughing response | 2 minutes after administration
  Grading based on the number and duration of coughs: Grade I, no coughing, breathing is even; Grade II, a single mild cough; Grade III, multiple coughs lasting less than 15 seconds; Grade IV, continuous coughing lasting more than 15 seconds
Blood pressure | before injection of Tegilidine or Sufentanil (T0), 2 minutes after injection (T1), 1 minute before intubation (T2), 1 minute after intubation (T3), and 3 minutes after intubation (T4）
  Blood pressure before and after administration, and before and after intubation
Heart rate | before injection of Tegilidine or Sufentanil (T0), 2 minutes after injection (T1), 1 minute before intubation (T2), 1 minute after intubation (T3), and 3 minutes after intubation (T4）
  heart rate before and after administration, and before and after intubation
Adverse reaction | 2 minutes after administration
  such as respiratory depression, vomiting, nausea, itching, etc.)

CONTACTS AND LOCATIONS:
Overall Officials: Xiaobao Zhang, Doctor, Study Director — Xuzhou Medical University Affiliated Hospital of Lianyungang: Lianyungang No 1 People's Hospital
Locations (1):
- The Affiliated Lianyungang Hospital of Xuzhou Medical University, Lianyungang, Jiangsu, China